CLINICAL TRIAL: NCT04093453
Title: The Acute Effect of Propionate on Energy Homeostasis
Acronym: PROEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18hh4373
Record Dates: First submitted 2019-08-05; First posted 2019-09-18 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-03

CONDITIONS: Obesity
Keywords: Short Chain Fatty Acids; Propionate; Energy Expenditure; Lipid Oxidation
MeSH Terms: conditions — Obesity | interventions — Sodium Chloride; Exercise; sodium propionate

STUDY DESIGN:
Intervention Model Description: This protocol consisted of three individual trials.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be masked to the contents of the capsules (sodium propionate or sodium chloride). They will not be masked to whether it is a resting or exercise or fasting condition as this is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo + Fasting (Placebo Comparator): Sodium Chloride tested in a fasting state. Participants will be fasting for duration of study visit (360 minutes).
  Interventions: Other: Placebo (Sodium Chloride)
- Placebo + Exercise (Placebo Comparator): Sodium Chloride tested in an exercise state. Participants will have the placebo then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Interventions: Other: Placebo (Sodium Chloride); Other: Exercise
- Placebo + Post-prandial (Placebo Comparator): Sodium Chloride tested in a post-prandial state. Participants will have the placebo then a mixed liquid meal test is given.
  Interventions: Other: Placebo (Sodium Chloride)
- Propionate and Fasting (Experimental): Sodium Propionate tested in a fasting state. Participants will be fasting for duration of study visit (360 minutes).
  Interventions: Dietary Supplement: Sodium Propionate
- Propionate and Exercise (Experimental): Sodium Propionate tested in an exercise state. Participants will have the sodium propionate then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Interventions: Other: Exercise; Dietary Supplement: Sodium Propionate
- Propionate and Post-prandial (Experimental): Sodium Propionate tested in a post-prandial state. Participants will have the sodium propionate then a mixed liquid meal test is given.
  Interventions: Dietary Supplement: Sodium Propionate

INTERVENTIONS:
Other: Placebo (Sodium Chloride) — Participant receive Placebo (Sodium Chloride)
  Arms: Placebo + Exercise; Placebo + Fasting; Placebo + Post-prandial
Other: Exercise — 1 hour exercise
  Arms: Placebo + Exercise; Propionate and Exercise
Dietary Supplement: Sodium Propionate — Participant receive Sodium Propionate
  Arms: Propionate and Exercise; Propionate and Fasting; Propionate and Post-prandial

SUMMARY:
The research project aims to examine the effect of a dietary supplement called propionate on how the human body in healthy adults aged (18- 65 years) responds to during fasting, exercise and following a liquid mixed meal test and how that would affect energy homeostasis and substrate oxidation.

DETAILED DESCRIPTION:
Dietary fibres have long been recognised for their important role in a healthy diet due to their negative association with, and even management of, chronic diseases such as obesity, diabetes, metabolic syndrome, cardiovascular disease and inflammatory-bowel disease among others.Emerging evidence has suggested that these benefits could largely be attributed to short chain fatty acids (SCFA) (acetate, propionate and butyrate), the main by-products of fibre fermentation in the gut. Previous research has demonstrated that a long-term elevation in the SCFA propionate significantly reduced body weight gain in overweight adults and reduced liver fat storage.

The current project will examine potential mechanisms for the positive effect of propionate on energy homeostasis and metabolic profile.The effects of propionate on circulating glucose, insulin, gut hormones and lipid levels at rest, following moderate-intensity exercise and mixed meal tolerance test will be examined.

To acutely increase propionate absorption from the gut the present project will use a simple nutritional supplement: sodium propionate in a hydroxypropylmethyl cellulose (HPMC) capsule. This capsule is coated with an enteric film which prevents gastric digestion until the capsule reaches the intestine. This nutritional supplement has been used in human volunteers in a previously approved ethics application (12/LO/1769: Oral propionate and glucose homeostasis). A 5g acute dose of sodium propionate had previously been tested and reported no adverse effects . The MHRA have confirmed that encapsulated sodium propionate is not classed as an investigative medicinal product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (body mass index (BMI) of 18-35 kg/m2)
* Age between 18-65 years (inclusive)

Exclusion Criteria:

* Weight change of ≥ 3kg in the preceding 2 months
* Current smokers
* Substance abuse
* Excess alcohol intake
* Pregnancy
* Diabetes
* Cardiovascular disease
* Cancer
* Gastrointestinal disease e.g. inflammatory bowel disease or irritable bowel syndrome
* Kidney disease
* Liver disease
* Pancreatitis
* Started new medication within the last 3 months likely to interfere with energy metabolism, appetite regulation and hormonal balance, including: anti-inflammatory drugs or steroids, antibiotics, androgens, phenytoin, erythromycin or thyroid hormones.
* Involved in current research or have recently been involved in any research prior to recruitment in the past 12 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chambers, PhD, Study Director — Imperial College London; Gary Frost, Professor, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 53 individual participants were enrolled in the entire study.
  25 enrolled in Fasted Study (all new). 25 enrolled in Postprandial Study (16 new, 9 had previously enrolled in Fasted study).
  25 enrolled in Exercise Study (12 new, 13 had previously enrolled in Fasted or Postprandial studies).
  The participant flow is therefore presented for the three individual study periods (25 starting each study period).
Groups:
- Fasted Study: Placebo/Propionate: Sodium Chloride tested in a fasted state. Participants will be fasting for duration of study visit (360 minutes).
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
  then
  Sodium Propionate tested in a fasted state. Participants will be fasting for duration of study visit (360 minutes).
  Propionate (Sodium Propionate): Participant receive Propionate (Sodium Propionate)
- Fasted Study: Propionate/Placebo: Sodium Propionate tested in a fasted state. Participants will be fasting for duration of study visit (360 minutes).
  Propionate (Sodium Propionate): Participant receive Propionate (Sodium Propionate)
  then
  Sodium Chloride tested in a fasted state. Participants will be fasting for duration of study visit (360 minutes).
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
- Post-Prandial Study: Placebo/Propionate: Sodium Chloride tested in a post-prandial state. Participants will have the placebo then a mixed liquid meal test is given.
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
  then
  Sodium Propionate tested in a post-prandial state. Participants will have the Propionate then a mixed liquid meal test is given.
  Propionate (Sodium Propionate): Participant receive Propionate (Sodium Propionate)
- Post-Prandial Study: Propionate/Placebo: Sodium Propionate tested in a post-prandial state. Participants will have the Propionate then a mixed liquid meal test is given.
  Propionate (Sodium Propionate): Participant receive Propionate (Sodium Propionate)
  then
  Sodium Chloride tested in a post-prandial state. Participants will have the placebo then a mixed liquid meal test is given.
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
- Exercise Study: Placebo/Propionate: Sodium Chloride tested in an exercise state. Participants will have the placebo then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride) Exercise: 1 hour exercise
  then
  Sodium Propionate tested in an exercise state. Participants will have the Propionate then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Propionate (Sodium Propionate): Participant receive Propionate (Sodium Propionate) Exercise: 1 hour exercise
- Exercise Study: Propionate/Placebo: Sodium Propionate tested in an exercise state. Participants will have the Propionate then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Propionate (Sodium Propionate): Participant receive Propionate (Sodium Propionate) Exercise: 1 hour exercise
  then
  Sodium Chloride tested in an exercise state. Participants will have the placebo then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride) Exercise: 1 hour exercise
Period: Fasted Study
Arm/Group | Fasted Study: Placebo/Propionate | Fasted Study: Propionate/Placebo | Post-Prandial Study: Placebo/Propionate | Post-Prandial Study: Propionate/Placebo | Exercise Study: Placebo/Propionate | Exercise Study: Propionate/Placebo
Started | 12 | 13 | 0 | 0 | 0 | 0
Completed | 10 | 9 | 0 | 0 | 0 | 0
Not Completed | 2 | 4 | 0 | 0 | 0 | 0
Period: Postprandial Study
Arm/Group | Fasted Study: Placebo/Propionate | Fasted Study: Propionate/Placebo | Post-Prandial Study: Placebo/Propionate | Post-Prandial Study: Propionate/Placebo | Exercise Study: Placebo/Propionate | Exercise Study: Propionate/Placebo
Started | 0 | 0 | 12 | 13 | 0 | 0
Completed | 0 | 0 | 9 | 11 | 0 | 0
Not Completed | 0 | 0 | 3 | 2 | 0 | 0
Period: Exercise Study
Arm/Group | Fasted Study: Placebo/Propionate | Fasted Study: Propionate/Placebo | Post-Prandial Study: Placebo/Propionate | Post-Prandial Study: Propionate/Placebo | Exercise Study: Placebo/Propionate | Exercise Study: Propionate/Placebo
Started | 0 | 0 | 0 | 0 | 13 | 12
Completed | 0 | 0 | 0 | 0 | 10 | 9
Not Completed | 0 | 0 | 0 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis of 'new' participants - first assigned study.
Groups:
- Fasted Study: Sodium Chloride tested in a fasting state. Participants will be fasting for duration of study visit (360 minutes).
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
  Theb
  Sodium Propionate tested in a fasting state. Participants will be fasting for duration of study visit (360 minutes).
  Sodium Propionate: Participant receive Sodium Propionate
- Post-prandial Study: Sodium Chloride tested in a post-prandial state. Participants will have the placebo then a mixed liquid meal test is given.
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
  Then
  Sodium Propionate tested in a post-prandial state. Participants will have the sodium propionate then a mixed liquid meal test is given.
- Exercise Study: Sodium Chloride tested in an exercise state. Participants will have the placebo then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
  Exercise: 1 hour exercise
  Then
  Sodium Propionate tested in an exercise state. Participants will have the sodium propionate then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Exercise: 1 hour exercise
  Sodium Propionate: Participant receive Sodium Propionate
- Total: Total of all reporting groups
Arm/Group | Fasted Study | Post-prandial Study | Exercise Study | Total
Number analyzed (Participants) | 25 | 16 | 12 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 16 | 12 | 53
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 4 | 23
  Male | 13 | 9 | 8 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25 | 16 | 12 | 53
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (0.7) | 24.7 (0.8) | 24.5 (0.7) | 24.1 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Resting Energy Expenditure
Description: Changes in Resting Energy Expenditure between sodium propionate and sodium chloride (control).
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: kcal/min
Arm/Group | Placebo + Fasting | Propionate and Fasting
Number analyzed (Participants) | 19 | 19
kcal/min | 1.013 (0.034) | 1.040 (0.039)

2. Primary Outcome: Changes in Resting Lipid Oxidation
Description: Changes in Resting Lipid Oxidation between sodium propionate and sodium chloride (control).
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: g/min
Arm/Group | Placebo + Fasting | Propionate and Fasting
Number analyzed (Participants) | 19 | 19
g/min | 0.032 (0.007) | 0.042 (0.007)

3. Primary Outcome: Changes in Energy Expenditure During Exercise
Description: Changes in Energy Expenditure between sodium propionate and sodium chloride (control) during exercise.
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: kcal/min
Arm/Group | Placebo + Exercise | Propionate and Exercise
Number analyzed (Participants) | 19 | 19
kcal/min | 5.085 (0.330) | 4.991 (0.328)

4. Primary Outcome: Changes in Lipid Oxidation During Exercise
Description: Changes in Lipid Oxidation between sodium propionate and sodium chloride (control) during exercise.
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: g/min
Arm/Group | Placebo + Exercise | Propionate and Exercise
Number analyzed (Participants) | 19 | 19
g/min | 0.284 (0.032) | 0.287 (0.030)

5. Primary Outcome: Changes in Energy Expenditure Post-prandially
Description: Changes in Energy Expenditure between sodium propionate and sodium chloride (control) post-prandially.
Time Frame: 300 minutes
Measure: Mean (Standard Deviation); unit: kcal/min
Arm/Group | Placebo + Post-prandial | Propionate and Post-prandial
Number analyzed (Participants) | 20 | 20
kcal/min | 1.057 (0.044) | 1.072 (0.046)

6. Primary Outcome: Changes in Lipid Oxidation Post-prandially
Description: Changes in Lipid Oxidation between sodium propionate and sodium chloride (control) post-prandially.
Time Frame: 300 minutes
Measure: Mean (Standard Deviation); unit: g/min
Arm/Group | Placebo + Post-prandial | Propionate and Post-prandial
Number analyzed (Participants) | 20 | 20
g/min | 0.027 (0.005) | 0.025 (0.005)

7. Primary Outcome: Changes in Glucose Concentrations Post-prandially
Description: Changes in glucose concentrations between sodium propionate and sodium chloride (control) post-prandially.
Time Frame: 300 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo + Post-prandial | Propionate and Post-prandial
Number analyzed (Participants) | 20 | 20
mmol/L | 5.38 (0.133) | 5.40 (0.141)

8. Primary Outcome: Changes in Glucose Concentrations During Exercise
Description: Changes in glucose concentrations between sodium propionate and sodium chloride (control) during exercise.
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo + Exercise | Propionate and Exercise
Number analyzed (Participants) | 19 | 19
mmol/L | 4.35 (0.09) | 4.47 (0.07)

9. Primary Outcome: Changes in Subjective Thirst Post-prandially Using a Visual Analog Scale (100 mm).
Description: Changes in subjective thirst between sodium propionate and sodium chloride (control) post-prandially. Volunteers completed the visual analog scale using a pen (Biro, black) with scales printed (Sharp MX-7580N ) on paper (A4, white). Visual analog scales were 100 mm in length. Minimum (0 mm) mean low subjective thirst. High (100 mm) mean high subjective thirst.
Time Frame: 300 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Post-prandial | Propionate and Post-prandial
Number analyzed (Participants) | 20 | 20
mm | 15.7 (4.3) | 14.5 (4.0)

10. Primary Outcome: Changes in Subjective Thirst During Exercise With Visual Analog Scales (100 mm)
Description: Changes in subjective thirst between sodium propionate and sodium chloride (control) during exercise. Volunteers completed the visual analog scale using a pen (Biro, black) with scales printed (Sharp MX-7580N ) on paper (A4, white). Visual analog scales were 100 mm in length. Minimum (0 mm) mean low subjective thirst. High (100 mm) mean high subjective thirst.
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Exercise | Propionate and Exercise
Number analyzed (Participants) | 19 | 19
mm | 39.8 (5.3) | 46.8 (5.4)

11. Primary Outcome: Changes in Subjective Nausea During Exercise With Visual Analog Scales (100 mm)
Description: Changes in subjective nausea between sodium propionate and sodium chloride (control) during exercise. Volunteers completed the visual analog scale using a pen (Biro, black) with scales printed (Sharp MX-7580N ) on paper (A4, white). Visual analog scales were 100 mm in length. Minimum (0 mm) mean low subjective nausea. High (100 mm) mean high subjective nausea.
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Exercise | Propionate and Exercise
Number analyzed (Participants) | 19 | 19
mm | 2.9 (1.1) | 6.7 (3.4)

12. Primary Outcome: Changes in Subjective Hunger During Exercise With Visual Analog Scales (100 mm)
Description: Changes in subjective hunger between sodium propionate and sodium chloride (control) during exercise. Volunteers completed the visual analog scale using a pen (Biro, black) with scales printed (Sharp MX-7580N ) on paper (A4, white). Visual analog scales were 100 mm in length. Minimum (0 mm) mean low subjective hunger. High (100 mm) mean high subjective hunger.
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Exercise | Propionate and Exercise
Number analyzed (Participants) | 19 | 19
mm | 51.7 (5.7) | 57.2 (5.3)

13. Secondary Outcome: Changes in GLP-1 Concentration
Description: Changes in GLP-1 concentrations between sodium propionate and sodium chloride (control) post-prandially.
Time Frame: 300 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Placebo + Postprandial: Sodium Chloride tested in a post-prandial state. Participants will have the placebo then a mixed liquid meal test is given.
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
- Propionate and Postprandial: Sodium Chloride tested in a post-prandial state. Participants will have the sodium propionate then a mixed liquid meal test is given.
  Sodium Propionate: Participant receive Sodium Propionate
Arm/Group | Placebo + Postprandial | Propionate and Postprandial
Number analyzed (Participants) | 20 | 20
mmol/L | 67.9 (7.1) | 70.5 (6.2)

14. Secondary Outcome: Changes in Insulin Concentration
Description: Changes in insulin concentrations between sodium propionate and sodium chloride (control) during fasting
Time Frame: 360 minutes
Measure: Mean (Standard Deviation); unit: μU/mL
Arm/Group | Placebo + Fasting | Propionate and Fasting
Number analyzed (Participants) | 19 | 19
μU/mL | 7.70 (0.48) | 7.87 (0.59)

15. Secondary Outcome: Changes in Glucose Concentration
Description: Changes in glucose concentrations between sodium propionate and sodium chloride (control) during fasting
Time Frame: 360 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo + Fasting | Propionate and Fasting
Number analyzed (Participants) | 19 | 19
mmol/L | 4.12 (0.08) | 4.14 (0.08)

16. Secondary Outcome: Changes in Free Fatty Acid Concentration
Description: Changes in free fatty acid concentrations between sodium propionate and sodium chloride (control) during fasting
Time Frame: 360 minutes
Population: Data not yet analysed.
Arm/Group | Placebo + Fasting | Propionate and Fasting
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Changes in Subjective Nausea With Visual Analog Scales (100 mm)
Description: Changes in subjective nausea between sodium propionate and sodium chloride (control) during fasting. Volunteers completed the visual analog scale using a pen (Biro, black) with scales printed (Sharp MX-7580N ) on paper (A4, white). Visual analog scales were 100 mm in length. Minimum (0 mm) mean low subjective nausea. High (100 mm) mean high subjective nausea.
Time Frame: 360 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Fasting | Propionate and Fasting
Number analyzed (Participants) | 19 | 19
mm | 48.0 (4.11) | 44.8 (5.25)

18. Secondary Outcome: Changes in Subjective Hunger With Visual Analog Scales (100 mm)
Description: Changes in subjective hunger between sodium propionate and sodium chloride (control) during fasting. Volunteers completed the visual analog scale using a pen (Biro, black) with scales printed (Sharp MX-7580N ) on paper (A4, white). Visual analog scales were 100 mm in length. Minimum (0 mm) mean low subjective hunger. High (100 mm) mean high subjective hunger.
Time Frame: 360 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Fasting | Propionate and Fasting
Number analyzed (Participants) | 19 | 19
mm | 48.0 (4.11) | 44.8 (5.25)

19. Secondary Outcome: Changes in Subjective Thirst Using Visual Analog Scales (100 mm)
Description: Changes in subjective thirst between sodium propionate and sodium chloride (control) during fasting. Volunteers completed the visual analog scale using a pen (Biro, black) with scales printed (Sharp MX-7580N ) on paper (A4, white). Visual analog scales were 100 mm in length. Minimum (0 mm) mean low subjective thirst. High (100 mm) mean high subjective thirst.
Time Frame: 360 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Fasting | Propionate and Fasting
Number analyzed (Participants) | 19 | 19
mm | 24.7 (5.43) | 23.2 (5.25)

20. Secondary Outcome: Changes in Insulin Concentration
Description: Changes in insulin concentrations between sodium propionate and sodium chloride (control) during exercise
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: μU/mL
Groups:
- Propionate and Exercise: Sodium Chloride tested in an exercise state. Participants will have the sodium propionate then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Placebo (Sodium Propionate): Participant receive Placebo (Sodium Propionate)
  Exercise: 1 hour exercise
Arm/Group | Placebo + Exercise | Propionate and Exercise
Number analyzed (Participants) | 19 | 19
μU/mL | 5.34 (0.39) | 5.63 (0.55)

21. Secondary Outcome: Changes in Insulin Concentration
Description: Changes in insulin concentrations between sodium propionate and sodium chloride (control) post-prandially.
Time Frame: 300 minutes
Measure: Mean (Standard Deviation); unit: μU/mL
Groups:
- Propionate and Postprandial: Sodium Propionate tested in a post-prandial state. Participants will have the sodium propionate then a mixed liquid meal test is given.
  Placebo (Sodium Propionate): Participant receive Sodium Propionate
Arm/Group | Placebo + Post-prandial | Propionate and Postprandial
Number analyzed (Participants) | 20 | 20
μU/mL | 29.88 (2.69) | 30.27 (2.17)

22. Secondary Outcome: Changes in Subjective Nausea Between Sodium Propionate and Sodium Chloride Post-prandially
Description: Changes in subjective nausea between sodium propionate and sodium chloride (control) post-prandially.
Time Frame: 300 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Postprandial | Propionate and Postprandial
Number analyzed (Participants) | 20 | 20
mm | 4.7 (1.8) | 5.3 (1.8)

23. Secondary Outcome: Changes in Subjective Hunger Between Sodium Propionate and Sodium Chloride Post-prandially With Visual Analog Scales (100 mm)
Description: Changes in subjective hunger between sodium propionate and sodium chloride (control) post-prandially. Volunteers completed the visual analog scale using a pen (Biro, black) with scales printed (Sharp MX-7580N ) on paper (A4, white). Visual analog scales were 100 mm in length. Minimum (0 mm) mean low subjective hunger. High (100 mm) mean high subjective hunger.
Time Frame: 300 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Postprandial | Propionate and Postprandial
Number analyzed (Participants) | 20 | 20
mm | 48.8 (5.0) | 43.7 (5.4)

ADVERSE EVENTS:
Time Frame: 2 years
Description: No adverse event observed or reported.
Groups:
- Placebo + Fasting Then Propionate and Fasting: Sodium Chloride tested in a fasting state. Participants will be fasting for duration of study visit (360 minutes).
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
  then
  Sodium Propionate tested in a fasting state. Participants will be fasting for duration of study visit (360 minutes).
  Sodium Propionate: Participant receive Sodium Propionate
- Placebo + Exercise Then Propionate and Exercise: Sodium Chloride tested in an exercise state. Participants will have the placebo then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
  Exercise: 1 hour exercise
  Then
  Sodium Propionate tested in an exercise state. Participants will have the sodium propionate then exercise will be performed at 40% of maximal aerobic capacity for one hour.
  Sodium Propionate: Participant receive Sodium Propionate.
  Exercise: 1 hour exercise
- Placebo + Postprandial Then Propionate and Postprandial: Sodium Chloride tested in a post-prandial state. Participants will have the placebo then a mixed liquid meal test is given.
  Placebo (Sodium Chloride): Participant receive Placebo (Sodium Chloride)
  Then
  Sodium Propionate tested in a post-prandial state. Participants will have the placebo then a mixed liquid meal test is given.
  Sodium Propionate: Participant receive Sodium Propionate
Arm/Group | Placebo + Fasting Then Propionate and Fasting | Placebo + Exercise Then Propionate and Exercise | Placebo + Postprandial Then Propionate and Postprandial
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT04093453/Prot_SAP_000.pdf